CLINICAL TRIAL: NCT03734809
Title: NEO-SPACE Trial: Neoadjuvant Pembrolizumab-Gemcitabine-Cisplatin Followed by Concurrent Pembrolizumab-Chemoradiation and Maintenance Pembrolizumab for Stage IVA Nasopharyngeal Cancer
Brief Title: NEO-SPACE Trial: Pembrolizumab and Chemoradiation in Nasopharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Edwin P Hui, Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC032
Record Dates: First submitted 2018-10-23; First posted 2018-11-08 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: NPC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pembrolizumab (Experimental): Total 51 weeks for 17 doses of pembrolizumab:
  * Neoadjuvant pembrolizumab-chemotherapy: 6 weeks (2 doses of pembrolizumab)
  * Concurrent pembrolizumab-chemoradiation: 9 weeks (3 doses of pembrolizumab
  * Maintenance pembrolizumab: 36 weeks (12 doses of pembrolizumab)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg every 3 weeks infusion
  Other Names: Concurrent Chemoradiation

SUMMARY:
This is an open label, single arm, non-randomized, multi-site, phase 2 clinical trial of neoadjuvant pembrolizumab in combination with gemcitabine-cisplatin for 2 cycles,followed by concurrent pembrolizumab-cisplain-radiation, and then maintainence pembrolizumab monotherpy given every 3 weeks for a total treatment duration of 12 months, in previously untreated stage IVA ( UICC 8 th Edition ) nasopharyngeal cancer(NPC).

DETAILED DESCRIPTION:
Nasopharyngeal cancer (NPC) is a predominantly Asian disease, with approximately 80% of the world's 86000 cases occurring in Asian countries (12). With advances in radiation technology such as intensity modulation radiotherapy (IMRT), local and nodal control exceeds 85-90% in most reported series. Distant metastasis remains the main mode of failure, particularly in locally advanced NPC. As an example, in a study by Pan et al (13), 5 years local and nodal control of 86% and 89% was achieved with concurrent chemo-IMRT respectively, but distant failure free survival of 77% and 72% was reported for patients with T4 and N3 disease respectively (AJCC 8th edition).

Current strategies to reduce distant metastasis, including the use of adjuvant chemotherapy have been inconclusive. One major disadvantage of adjuvant chemotherapy following the completion of chemoradiation is that approximately half of patients are unable to complete the full 3 cycles of adjuvant chemotherapy, due to treatment related toxicities. The use of induction chemotherapy has two potential benefits: the first is to downsize the tumour, making radiotherapy more tolerable; the second, it allows for patients to be able to complete the chemotherapy before the onset of chemoradiation associated toxicities.

There are at least two studies now supporting the use of induction chemotherapy. A recent publication by Ma et al (14), showed the addition of induction docetaxel, cisplatin and fluorouracil prior to concurrent chemoradiation resulted in 8% improvement (80% vs 72%) in 3-year failure-free survival. Similarly, Cao et al showed that 2 cycles of cisplatin and fluorouracil prior to chemoradiation improved the 3 years disease free survival in patients (15).

Gemcitabine and cisplatin has been shown to be more effective than 5-FU plus cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (16). There are currently no studies looking at the addition of anti-PD-1 monoclonal antibody such as pembrolizumab either in the in the induction or maintenance setting. Hence, we are proposing the use of pembrolizumab in combination with 2 cycles of gemcitabine and cisplatin chemotherapy followed by concurrent chemoradiation. Following completion of chemoradiation, patients will receive maintenance pembrolizumab for total treatment duration of one year. The main objective of this Phase II study is to test the safety, efficacy and tolerability of this combination in the setting of locally advanced NPC (limited to T4 or N3, stage IVA by UICC 8th edition), as this group has the greatest risk of recurrence after the current standard treatment.

Preliminary evidence supporting the clinical efficacy of pembrolizumab monotherapy in NPC came from the KEYNOTE-028 trial, which was a global, nonrandomized, multi-cohort, phase Ib trial of pembrolizumab in patients with PD-L1-positive advanced solid tumors (17). Key eligibility criteria for the NPC cohort included unresectable or metastatic disease, failure on prior standard therapy, and PD-L1 expression in 1% or more of tumor cells or tumor-infiltrating lymphocytes. Patients received pembrolizumab 10 mg/kg every 2 weeks up to 2 years or until disease progression or unacceptable toxicity. In the initial report, twenty-seven NPC patients was evaluated. Median age was 52.0 years (range, 18 to 68 years); 92.6% received prior therapies for recurrent or metastatic NPC; 70.4% had received three or more therapies. Partial response and stable disease were observed in seven and 14 patients, respectively, for an ORR of 25.9% (95% CI, 11.1 to 46.3) over a median follow-up of 20 months. Drug-related adverse events that occurred in 15% or more of patients included rash (25.9%), pruritus (25.9%), pain (22.2%), hypothyroidism (18.5%), and fatigue (18.5%). Grade ≥ 3 drug-related adverse events occurred in eight patients (29.6%), and there was one drug-related death (sepsis). It was concluded that pembrolizumab demonstrated antitumor activity and a manageable safety profile in patients with recurrent or metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of nasopharyngeal carcinoma (from primary lesion and/or lymph nodes) of WHO type II-III histology type will be enrolled in this study.
2. Tumor confirmed EBV positive by EBER ISH assay
3. AJCC 8th edition Stage IVA (i.e any T4 or any N3) based on the following diagnostic workup:

   1. Evaluation of tumor extent with MRI of the nasopharynx and neck. If MRI is medically contraindicated, CT scan with

      ≤ 3 mm and intravenous contrast is acceptable.
   2. Distant metastasis staging:

   i. CT scan with contrast of the chest, abdomen, and pelvis or a total body PET/CT scan; ii. Bone scan, if a PET/CT scan is not performed.
4. A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days plus an additional 120 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose after the last dose of study treatment and refrain from donating sperm during this period.
5. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
9. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to first dosing (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received any prior systemic anti-cancer therapy including investigational agents.
4. Has received any prior radiotherapy.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Subjects who have been treated and now have a viral load that is undetectable are eligible.
15. Has a known history of active TB (Bacillus Tuberculosis).
16. Has prior solid organ transplant or bone marrow transplant.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong
- National Cancer Centre of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Total 51 weeks for 17 doses of pembrolizumab:
  * Neoadjuvant pembrolizumab-chemotherapy: 6 weeks (2 doses of pembrolizumab)
  * Concurrent pembrolizumab-chemoradiation: 9 weeks (3 doses of pembrolizumab
  * Maintenance pembrolizumab: 36 weeks (12 doses of pembrolizumab)
  Pembrolizumab: 200mg every 3 weeks infusion
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 43
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 14
  Hong Kong | 29

OUTCOME MEASURES:

1. Primary Outcome: Two-year Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1), including
  * Increase in the sum of diameters of target lesion(s) identified at baseline to ≥ 20% and ≥ 5 mm from nadir
  * Unequivocal progression of non-target lesion(s) identified at baseline
  * Development of new lesion(s)
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants | 73.8 [60.5 to 87.1]

2. Secondary Outcome: Grade 4 Mucositis/Skin Reaction or Any Grade 5 Adverse Event Assessed to be Definitely, Probably, or Possibly Related to Protocol Treatment During the First Year
Description: use toxicity chart to capture
Time Frame: during the first year
Measure: Number; unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
participants | 0

3. Secondary Outcome: Grade 4 Mucositis/Skin Reaction or Any Grade 5 Adverse Event Assessed to be Definitely, Probably, or Possibly Related to Protocol Treatment Occurring After the First Year
Time Frame: after the first year, up to 24 months
Measure: Number; unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
participants | 0

4. Secondary Outcome: Patient Tolerability to Each Component (Neoadjuvant, Concurrent and Maintenance Part) of the Protocol Treatment Regimen
Time Frame: 2 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  Chemotherapy - neoadjuvant phase | 98.0
  Chemotherapy - Concurrent phase | 73.1
  Immunotherapy - neoadjuvant phase | 100.0
  Immunotherapy - Concurrent phase | 78.3
  Immunotherapy - maintenance phase | 78.1
  Radiotherapy | 100.0

5. Secondary Outcome: Other ≥ Grade 3 Adverse Events
Time Frame: 2 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  Dysphagia | 32.4
  Mucositis | 29.7
  Neutropenia | 29.7
  Radiation dermatitis | 24.3
  Anemia | 18.9
  Hyponatremia | 13.5
  Thrombocytopenia | 10.8

6. Secondary Outcome: Death During or Within 30 Days of Discontinuation of Protocol Treatment
Time Frame: during or within 30 days
Measure: Number; unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
participants | 0

7. Secondary Outcome: One- and Two-year Distant Metastases Rates
Time Frame: 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  One-year rate of distant metastases | 95.2 [88.8 to 100.0]
  Two-year rate of distant metastases | 83.0 [71.0 to 95.0]

8. Secondary Outcome: One- and Two-year Local-regional Progression Rates
Time Frame: 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  One-year rate of local-regional progression | 95.3 [88.9 to 100.0]
  Two-year rate of local-regional progression | 90.4 [81.5 to 99.3]

9. Secondary Outcome: One- and Two-year Rates of Second Primary Cancer
Time Frame: 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  One-year rate of secondary primary | 100.0 [100.0 to 100.0]
  Two-year rate of secondary primary | 97.5 [92.6 to 100]

10. Secondary Outcome: One- and Two-year Overall Survival Rates
Time Frame: 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 43
percentage of participants
  One-year rate of overall survival | 97.6 [93.0 to 100.0]
  Two-year rate of overall survivial | 92.9 [85.1 to 100.0]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 8/43
Serious Adverse Events (participants affected / at risk) | 17/43
Other Adverse Events (participants affected / at risk) | 32/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=43)
Fever (General disorders) | 6
Dysphagia (Gastrointestinal disorders) | 3
Infections and infestations - Other (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Sepsis (Immune system disorders) | 1
Alkaline phosphataseincrease (Gastrointestinal disorders) | 1
Relapse of mania (Psychiatric disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypothermia (General disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Thromboembolic event - Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Neck edema (General disorders) | 1
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=43)
Dysphagia (Gastrointestinal disorders) | 14
Mucositis (Gastrointestinal disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 13
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 10
Anemia (Blood and lymphatic system disorders) | 8
Hyponatremia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03734809/Prot_SAP_000.pdf